CLINICAL TRIAL: NCT05599659
Title: The Calgary Movement Disorders Advanced Care Pilot Program
Acronym: ACT for PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Veronica Bruno, MD, MPH, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: REB22-0545
Record Dates: First submitted 2022-10-12; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Parkinson's Disease and Parkinsonism
Keywords: Palliative Care
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: The clinical trial is a prospective cohort study analysing the effect of palliative care interventions on quality of life, patient satisfaction, carepartner burden and health care utilization patterns in patients living with parkisonism and their carepartners.
  Participants will:
  * Receive multidisciplinary palliative care.
  * Answer questions related to the quality of life, patient satisfaction, carepartner burden and health care utilization patterns.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Palliative care (Experimental): Participants will receive palliative care.
  Interventions: Behavioral: Palliative care

INTERVENTIONS:
Behavioral: Palliative care — It is a pilot model of outpatient clinical care for patients in advanced stages of PDRD that will allow earlier access to PC in this population. PC visits will be in person or by telemedicine every three months and complemented with phone calls by different team members when needed as defined by the PC team.
  The typical visit duration will be 2 to 2.5 hours and address nonmotor symptoms, goals of care, anticipatory guidance, difficult emotions, and carepartner support. Providers will communicate in-person or via notes during the clinic visit to increase interdisciplinary coordination and meet at the end of the day for discussion including follow-up plans.
  The team will consist of a neurologist, a registered nurse with palliative care experience and training, a psychology counselor, a social worker, spiritual counselor and a research assistant.
  Other Names: Advanced care

SUMMARY:
The goal of this clinical trial is to analyse the effect of palliative care interventions on quality of life, patient satisfaction, carepartner burden and health care utilization patterns in patients living with parkisonism and their carepartners.

Participants will:

* Receive multidisciplinary palliative care.
* Answer questions related to the quality of life, patient satisfaction, carepartner burden and health care utilization patterns.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have a PD diagnosis or another PDRD diagnosis (multiple system atrophy, corticobasal degeneration, progressive supranuclear palsy, or Lewy body dementia)
* Participants who have moderate to high PC needs based on the Palliative Care Needs Assessment Tool (PC-NAT)
* Participants who are between 20 and 100 years old

Exclusion Criteria:

* Immediate and urgent palliative care needs. These patients will be offered appropriate services immediately
* Participants who have other illnesses that could require PC e.g. metastatic cancer
* Participants already receiving PC and/or hospice
* Patients with a diagnosis of severe cognitive impairment (Montreal Cognitive Assessment <10). These patients will be offered appropriate services. Care partners can participate.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-04 (Estimated); Primary Completion 2024-11-04 (Estimated); Study Completion 2024-11-04 (Estimated)

PRIMARY OUTCOMES:
Changes in Quality of Life Alzheimer's Disease (QOL-AD) | Every 3 months for 2 years
  The QOL-AD is a 13-item questionnaire designed to provide both a patient and a caregiver report of the quality of life (QOL), it uses a scale of 1-4 (poor, fair, good, or excellent) to rate a variety of life domains, including the patient's physical health, mood, relationships, activities, and ability to complete tasks.
Changes in 12-Item Zarit Burden Interview (ZBI-12) | Every 3 months for 2 years
  ZBI-12 is validated as a screening tool for advanced illness. The ZBI-12 is rated on a 12 items scale, with the severity of burden using a range of responses from 0 to 4 points per item and a total score range of 0 to 48. Scoring 0-10 is considered as a no to mild burden; 10-20, a mild to moderate burden and >20, a high burden. It measures changes in physical, emotional, social, and financial problems that can be experienced by family caregivers.
Changes in Health Care Utilization survey | Every 3 months for 2 years
  We will perform a Health Service Utilization Survey to measure changes in the number of hospitalizations, emergency room visits, home health services, and nursing home placement.

SECONDARY OUTCOMES:
Changes in Edmonton Symptom Assessment Scale revised for Parkinson's Disease (ESAS-PD) | Every 3 months for 2 years
  The ESAS is a comprehensive, yet brief and practical self-reporting tool of symptom severity (intensity) for nine common symptoms of advanced cancer (pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being, shortness of breath), with the option of adding a tenth patient-specific symptom. It rates the severity of each symptom on a 0 to 10 scale, where 0 represents the absence (or best possible intensity) of the symptom and 10 represents the worst possible severity.
Changes in the Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being (FACIT- Sp-12) | Every 3 months for 2 years
  The 12-item Spiritual Well-Being Scale (FACIT-Sp-12) is the most widely used measure of spiritual well-being among those with long-term illness. The FACIT-Sp comprises 12 statements, or items, each of which is rated on a 5-point scale by the respondent based on how true the item was during the past week, 0 for not at all, 1 for a little bit, 2 for somewhat, 3 for quite a bit and 5 for very much.
Semi-structured Qualitative Interview to receive Patient and Care Partner recommendations | Every 3 months for 2 years
  It will be performed on patients and care partners for optimizing the palliative care services provided and delivery methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Movement Disorder Program, Foothills Medical Center, Alberta Health Services, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No